CLINICAL TRIAL: NCT06142357
Title: Prospective Observational Study With Retrospective Part to Evaluate Secukinumab Drug Survival, Effectiveness and Tolerability in Pediatric Patients With Moderate-to-severe Plaque Psoriasis
Brief Title: Secukinumab Drug Survival, Effectiveness and Tolerability in Pediatric Patients With Psoriasis
Acronym: SPARROW
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457LRU01
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Moderate-to-severe Plaque Psoriasis
Keywords: Secukinumab,; psoriasis,; pediatric patients,; NIS
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Secukinumab: Pediatric patients with moderate-to-severe plaque psoriasis receiving secukinumab.
  Interventions: Other: Secukinumab

INTERVENTIONS:
Other: Secukinumab — There is no treatment allocation. Patients administered secukinumab by prescription will be enrolled
  Other Names: Cosentyx

SUMMARY:
Multicenter, non-interventional, cohort study in pediatric patients with moderate to severe plaque-type psoriasis. Retrospective data collection is planned at patients' inclusion.

DETAILED DESCRIPTION:
This observational study will be performed at healthcare facilities treating pediatric psoriasis patients. The study population will consist of a representative group of pediatric patients with moderate-to-severe plaque psoriasis for whom routine treatment with secukinumab according to the approved national label is initiated during 4 to 16 weeks Retrospective data collection is planned at patients' inclusion. Prospective data collection will continue during follow-up routine visits until secukinumab discontinuation or maximum duration of follow-up for 104 weeks after index date.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and legal representative's permission for study participation obtained prior to beginning of participation in the study.
2. Age ≥6 to <18 years old.
3. Established diagnosis of active moderate-to-severe plaque psoriasis defined as a PASI score ≥ 10, body surface area (BSA) involvement of ≥10% and PGA score ≥ 3 only or with concomitant psoriatic arthritis.
4. Failure or intolerance of prior psoriasis treatment.
5. Patient was prescribed with secukinumab within 4-16 weeks before inclusion.
6. Decision for secukinumab prescription was made by the attending physician according to the approved national label during routine clinical practice, regardless of this non-interventional study conduct.

Exclusion Criteria:

1. Known or suspected severe hypersensitivity for secukinumab, formulation excipients, or injection device components (i.e., latex).
2. History of chronic recurrent infection.
3. Clinically significant infection exacerbation, including active tuberculosis.
4. Age <6 years or ≥18 years.
5. Pregnancy and breastfeeding.
6. Patients participating in parallel in an interventional clinical trial.
7. Patients participating in parallel in other Novartis-sponsored non-interventional study generating primary data for secukinumab.
8. Patients within the safety follow-up phase of interventional study.
9. Active inflammatory bowel disease at inclusion.
10. Patients who received any vaccine within 4 weeks prior to secukinumab initiation.
11. Any medical or psychological condition in the investigator's opinion which may prevent the study participation.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients aged ≥6 to <18 years old with moderate-to-severe plaque psoriasis after failure/intolerance of frontline treatment in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Drug survival rate of secukinumab | 52 weeks
  Drug survival is defined as time from the index date (defined as secukinumab treatment initiation) until discontinuation of secukinumab (defined as ≥2 missed consecutive doses with drug discontinuation proved by investigator in eCRF).

SECONDARY OUTCOMES:
Secukinumab survival rates | Week 24, week 52, and week 104 after the index date
  Secukinumab survival rate is defined as proportion of patients who have not discontinued treatment due to reasons other than lack of efficacy.
Time to treatment discontinuation due to ineffectiveness | Week 12, week 24, week 52, week 104
  Time from index date to treatment discontinuation due to ineffectiveness
Proportion of patients achieving PASI 75 responses | Baseline (study inclusion), week 24, week 52, and week 104 after the index date
  Psoriasis Area and Severity Index (PASI) takes into account the extent of the disease, as well as the severity of erythema, scaling, and thickness in different body areas affected by psoriasis.
  A PASI 75 represents an improvement in the PASI score of at least 75% as compared with baseline.
Proportion of patients achieving PASI 90 responses | Baseline (study inclusion), week 24, week 52, and week 104 after the index date
  Psoriasis Area and Severity Index (PASI) takes into account the extent of the disease, as well as the severity of erythema, scaling, and thickness in different body areas affected by psoriasis.
  A PASI 90 represents an improvement in the PASI score of at least 90% as compared with baseline.
Proportion of patients achieving PASI 100 responses | Baseline (study inclusion), week 24, week 52, and week 104 after the index date
  Psoriasis Area and Severity Index (PASI) takes into account the extent of the disease, as well as the severity of erythema, scaling, and thickness in different body areas affected by psoriasis.
  A PASI 100 response corresponds to complete clearing of psoriasis (PASI = 0).
Proportion of patients achieving a physicians' global assessment (PGA) 0/1 response | Baseline (study inclusion), week 24, week 52, and week 104 after the index date
  Proportion of patients achieving a physicians' global assessment 0/1 response: clear/almost clear skin
Adverse events (AEs) of special interest | Week 12, week 24, week 52, week 104 after the index date
  Adverse events (AEs) of special interest:
  Inflammatory Bowel Disease, malignancy, tuberculosis, serious infections, candidiasis, acute injection site reaction, immunogenicity
Proportion of patients discontinued secukinumab by reason | Week 12, week 24, week 52 and week 104
  Proportion of patients discontinued secukinumab by reason:
  * Lack of efficacy
  * Adverse events
  * Administrative reasons (no medication available in the hospital, etc.)
  * Lack of patient's adherence
  * Patient's or legal representative's wish
  * Other
Drug survival rate | 104 weeks
  Drug survival is defined as time from the index date (defined as secukinumab treatment initiation) until discontinuation of secukinumab (defined as ≥2 missed consecutive doses with drug discontinuation proved by investigator in eCRF).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Russia (13):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Grozny
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Mytishchi
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Tolyatti
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yakutsk

IPD SHARING:
Plan to Share IPD: No